CLINICAL TRIAL: NCT00005249
Title: Epidemiology of Blood Pressure, Insulin, Salt Transport
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1131; R01HL039748 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity

SUMMARY:
To determine the roles of insulin, lipids, body weight and ion transport in blood pressure regulation.

DETAILED DESCRIPTION:
BACKGROUND:

Insulin levels are consistently related to blood pressure, obesity, and blood lipids. Insulin level correlation with sodium-lithium countertransport is limited to only one available study done in white, normotensive, predominantly normal weight women aged 45-52. The relationship between cellular sodium-hydrogen exchange activity and hypertension has been studied in rats and in a small study in humans. Correlation of this transport with weight, fasting insulin and lipid levels, and sodium-lithium countertransport was not available in 1989.

DESIGN NARRATIVE:

The study was cross-sectional. Subjects were stratified by weight: plus or minus 10 percent of desirable weight; 11 to 30 percent over desirable weight; and 30 percent over desirable weight; and by diastolic blood pressure: 80; 80-89; 90-99 mmHg. Blood pressure, height, weight, waist and hip girth, skinfold, fasting and post-glucose load insulin, glucose, lipids, creatinine, maximal rates of red blood cell sodium-lithium countertransport and platelet sodium-hydrogen exchange, pH, and calcium concentrations were measured. The strength and independence among these continuous variables were measured by Pearson correlations, partial correlations, and multiple regressions within each stratum, and if appropriate, over all strata. The study examined the hypotheses that: part of the relationship between obesity and blood pressure was due to insulin effects and/or lipid effects on ion transport; the relationship between ion transport and blood pressure was related to an abnormality of sodium-hydrogen exchange, for which the observed increase in sodium-lithium countertransport was a marker; increased blood pressure was related to the alteration of intracellular pH and/or calcium concentration.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-09; Study Completion 1991-08 (Actual)

REFERENCES:
- [Background] Bunker CH, Wing RR, Becker DJ, Kuller LH. Sodium-lithium countertransport activity is decreased after weight loss in healthy obese men. Metabolism. 1993 Aug;42(8):1052-8. doi: 10.1016/0026-0495(93)90022-g. PMID 8345810